CLINICAL TRIAL: NCT02031692
Title: Efficacy of Vitamin D and Calcium Supplementation on the Prevention of Recurrences in Benign Paroxysmal Positional Vertigo: A Prospective Multicenter Randomized Trial
Brief Title: Efficacy of Vitamin D and Calcium Supplementation on the Prevention of Recurrences in BPPV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Ji-Soo Kim, Professor and Chairman, Department of Neurology, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-2013-092; HI10C2020 (Other Grant/Funding Number: Ministry of Health and Welfare); 1386-5650-7389-0156 (Other: Ministry of Food and Drug Safety, Korea)
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: Benign paroxysmal positional vertigo; Vitamin D; Calcium; Prevention
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo | interventions — Cholecalciferol; Calcium; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D and calcium supplement (Active Comparator)
  Interventions: Drug: 400IU cholecalciferol and 500mg of elemental calcium as calcium carbonate
- Control (No Intervention)

INTERVENTIONS:
Drug: 400IU cholecalciferol and 500mg of elemental calcium as calcium carbonate — The patients allocated to the intervention group will have a test for serum vitamin D, and receive 800 IU of vitamin D and 1000 mg of calcium as calcium carbonate when the serum vitamin D is decreased. The patients in the control group will be followed up without intervention for one year.
  Other Names: CAVID CHEWABLE TAB, Takeda Pharmaceuticals
  Arms: Vitamin D and calcium supplement

SUMMARY:
The purpose of this study is to determine whether the supplementation of vitamin D and calcium prevents recurrences of benign paroxysmal positional vertigo in patients with vitamin D deficiency/insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* brief episodes of vertigo induced by head motion
* a typical positioning nystagmus characteristic of BPPV
* no supplementation of vitamin D or calcium at the time of recruitment
* informed consent to participate in this study
* subject treated by repositioning maneuver

Exclusion Criteria:

* other identifiable disorders of the central nervous system
* supplementation of vitamin D or calcium at the time of recruitment
* pregnancy
* a history of an allergic reaction, or a medically significant adverse reaction to the investigational product
* contraindication to cholecalciferol and calcium carbonate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2013-12; Primary Completion 2017-05-26 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Recurrence frequency of benign paroxysmal positional vertigo | Up to 1 year
  The intervention group will receive tablets containing 400IU cholecalciferol and 500mg of elemental calcium as calcium carbonate twice daily (CAVID CHEWABLE TAB, Takeda Pharmaceuticals) for 12 months when the initial serum vitamin D is decreased. The compliance will be determined by the percentage of consumed tablets from the delivered tablets during the follow-up period. Discontinuation of the supplementation due to adverse effects or other reasons will be registered using the telephone interview together with the primary outcome date. Participants in the control group will not have any intervention or placebo. They will not be allowed to take vitamin D or calcium as supplements during the follow-up. The primary outcome measure is the recurrence of BPPV after one year. Data on recurrences will be collected using a monthly telephone interview, and the patients will be asked to visit the clinic whenever they have the symptoms of BPPV. All the recurrences of BPPV will be included.

SECONDARY OUTCOMES:
Changes in serum 25-hydroxy vitamin D level | Up to 1 year
  In intervention group, the baseline vitamin D status of participants will be checked. And the level of 25-hydroxyvitamin D level will be rechecked at 2 months from the recruitment and at the end of the follow-up.
Falling frequency | Up to year
  To determine the supplementation of the vitamin D and calcium carbonate is effective to decrease falling frequency.
Fracture frequency | Up to 1 year
  To determine the supplementation of the vitamin D and calcium carbonate is effective to decrease fracture frequency.
Quality of life | Up to 1 year
  To determine the supplementation of the vitamin D and calcium carbonate is related to quality of life using UCLA-dizziness questionnaire
Recurrence rate of benign paroxysmal positional vertigo | Up to 1 year
  The intervention group will receive tablets containing 400IU cholecalciferol and 500mg of elemental calcium as calcium carbonate twice daily (CAVID CHEWABLE TAB, Takeda Pharmaceuticals) for 12 months when the initial serum vitamin D is decreased. The compliance will be determined by the percentage of consumed tablets from the delivered tablets during the follow-up period. Discontinuation of the supplementation due to adverse effects or other reasons will be registered using the telephone interview together with the primary outcome date. Participants in the control group will not have any intervention or placebo. They will not be allowed to take vitamin D or calcium as supplements during the follow-up. The primary outcome measure is the recurrence rate of BPPV after one year. Data on recurrences will be collected using a monthly telephone interview, and the patients will be asked to visit the clinic whenever they have the symptoms of BPPV. All the recurrences of BPPV will be included.

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Soo Kim, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National Universtiy Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Jeong SH, Kim JS, Shin JW, Kim S, Lee H, Lee AY, Kim JM, Jo H, Song J, Ghim Y. Decreased serum vitamin D in idiopathic benign paroxysmal positional vertigo. J Neurol. 2013 Mar;260(3):832-8. doi: 10.1007/s00415-012-6712-2. Epub 2012 Oct 25. PMID 23096068
- [Background] Jeong SH, Choi SH, Kim JY, Koo JW, Kim HJ, Kim JS. Osteopenia and osteoporosis in idiopathic benign positional vertigo. Neurology. 2009 Mar 24;72(12):1069-76. doi: 10.1212/01.wnl.0000345016.33983.e0. PMID 19307540
- [Derived] Jeong SH, Kim JS. Impaired Calcium Metabolism in Benign Paroxysmal Positional Vertigo: A Topical Review. J Neurol Phys Ther. 2019 Apr;43 Suppl 2:S37-S41. doi: 10.1097/NPT.0000000000000273. PMID 30883492